CLINICAL TRIAL: NCT05305183
Title: A Randomized, Double-blinded, Active-controlled, Multicentered Phase III Trial to Assess the Efficacy and Safety of Minodronate Tablets in Postmenopausal Women With Osteoporosis
Brief Title: A Phase III Clinical Study of Minodronate Tablets in Postmenopausal Women With Osteoporosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTP-MNLS-T-Ⅲ
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — YM 529

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alendronate Sodium Tablets and Minodronate Tablets -matching placebo (Active Comparator): subjects received 70 mg alendronate sodium tablet weekly and a minodronate tablet matching placebo monthly for 48 weeks.
  Interventions: Drug: Minodronate Tablets and Alendronate Sodium Tablets-matching placebo;Alendronate Sodium Tablets and Minodronate Tablets -matching placebo
- Minodronate Tablets and Alendronate Sodium Tablets-matching placebo (Experimental): subjects received 50mg minodronate tablets monthly and an alendronate sodium tablets -matching placebo weekly for 48 weeks.
  Interventions: Drug: Minodronate Tablets and Alendronate Sodium Tablets-matching placebo;Alendronate Sodium Tablets and Minodronate Tablets -matching placebo

INTERVENTIONS:
Drug: Minodronate Tablets and Alendronate Sodium Tablets-matching placebo;Alendronate Sodium Tablets and Minodronate Tablets -matching placebo — all subjects will receive Calcium Carbonate and Vitamin D3 Tablets as basic medication.

SUMMARY:
In the randomized, active-controlled, double-blinded, multicenter study, the efficacy and safety of monthly oral minodronate were examined and compared to that of weekly oral alendronate.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 46-80 years, menopause for more than 1 year, free to move，Estradiol ≤20pg/mL and follicle stimulating hormone ≥40IU/L in patients with simple hysterectomy;
2. Body mass index (BMI) is 18.5-30.0kg/m2, including critical value, BMI= weight (kg)/height 2 (m2);
3. Based on dual energy X-ray absorption (DXA)Determination, bone density (BMD) determination of lumbar vertebrae L1-L4 (At least 2 consecutive lumbar vertebrae for accurate measurement of BMD ) mean T ≤ -2.5SD, or T≤ -2.5SD on either side of the double hip femoral neck;
4. Understand the procedures and methods of this clinical study, voluntarily participate in and sign the informed consent form.

Exclusion Criteria:

1. Patients with conditions that affect BMD measurement, such as severe scoliosis or any lumbar L1-L4 fracture or hip fracture;
2. Patients with secondary osteoporosis;
3. Endocrine diseases or other diseases affecting bone metabolism that the investigator considers inappropriate, such as gonads, adrenal glands, primary parathyroid dysfunction, or malformed osteitis (Paget's bone disease), nephrotic rickets, osteomalacia, rheumatoid arthritis, osteogenesis imperfecta , poorly controlled hyperthyroidism or hypothyroidism;
4. Patients with serious primary diseases such as cardiovascular, cerebrovascular and hematopoietic system, and mental or nervous system diseases;
5. Patients with abnormal blood calcium: serum calcium or serum calcium corrected by albumin ≤2.0mmol/L or ≥2.9mmol/L;
6. Parathyroid hormone > 1.5 times the upper limit of normal;
7. Patients with severe gastrointestinal absorption dysfunction such as dysphagia, esophagitis, enteritis or peptic ulcer，crohn's disease and chronic pancreatitis;
8. Patients with delayed obstruction of the esophagus, such as narrow or loose esophagus;
9. patients has previous or co-existing malignancies (except skin basal cell carcinoma and carcinoma in situ of the cervix, which have been cured for more than 3 years);
10. The patient who are deformed, disabled, unable to work or in a critical condition; which difficult to evaluate the effectiveness and safety of drugs accurately ;
11. Patients with type 1 diabetes or type 2 diabetes with poor glycemic control and severe acute and chronic complications;
12. Patients had received any other investigational drug/device treatment within 3 months prior to enrollment;
13. Patients with renal insufficiency or severe renal impairment(Ccr<35mL/min);
14. Patients with abnormal liver function (ALT or AST≥2.0 times the upper limit of normal);
15. Allergic constitution or allergic to study related drugs (calcium, vitamin D, minodronic acid or similar drugs);
16. Hepatitis B surface antigen (HBsAg) positive or hepatitis B core antibody (HBcAb) positive with HBV-DNA positive, hepatitis C virus (HCV) antibody positive with HCV-RNA positive, human immunodeficiency virus (HIV) positive, syphilis antibody positive;
17. The patients has previous or co-existing osteomyelitis or osteonecrosis of the mandible, the patients have dental surgery such as tooth extraction during the first 2 months of enrollment or during the trial;
18. The patients with a history of drug abuse or alcohol abuse within 6 months prior to enrollment;
19. The patients used the following drugs before enrollment: used oral bisphosphonate more than 3 months within 1 year or the cumulative use of oral bisphosphonate more than 1 year; used desomumab within 1 year;used intravenous bisphosphonate within the past 5 years;patients daily used systemic corticosteroid equivalent to prednisone > 5mg more than 14 days within 2 months (local external use is excluded) ;used calcitonin or active vitamin D complex within 6 weeks; used selective estrogen receptor modulators or estrogen replacement therapy for more than 1 month within 6 months;Qianggu capsule, total flavone of Epimedium, Jintiange capsule, Xianling Gubao capsule, Qigu capsule, Gushukang capsule and Zuogui pill were used for more than 3 months in 6 months;
20. Other patients that the investigator believes are not suitable for enrollment.

Ages: 46 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
The average rate of bone mineral density change of lumbar spine (L1-L4 ) was compared between 48 weeks after administration and before administration .the group of minodronate were examined and compared to that of alendronate. | 48 weeks

SECONDARY OUTCOMES:
The average rate of bone mineral density change of lumbar spine (L1-L4 ) was compared between 24 weeks after administration and before administration . | 24weeks
The change rate of bone turnover markers from baseline to 12、24、48 weeks, including serum type I collagen amino terminal peptide(P1NP) and serum C-terminal telopeptide of type 1 collagen (S-CTX ). | 12、24、48 weeks,
the change rates of bone density at the femoral neck and the whole hip from baseline to the end of 24 and 48 weeks. | 24、48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong New Time Pharmaceutical Co., LTD, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided